CLINICAL TRIAL: NCT03884972
Title: A Phase I/Ib Pilot Study of Combined Trabectedin and Venetoclax in Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma Resistant or Intolerant to a BTK Inhibitor
Brief Title: Trabectedin and Venetoclax in Treating Patients With Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma Resistant or Intolerant to a BTK Inhibitor
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Request by sponsor due to no enrollment of participants on study
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0302; NCI-2019-01555 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0302 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Refractory Chronic Lymphocytic Leukemia; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Trabectedin; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort I (BTK-refractory) (Experimental): Patients receive venetoclax PO QD beginning on day 1 for 5 weeks (cycle 1). Beginning in cycle 2, patients receive venetoclax PO QD and trabectedin IV over 3 hours on day 1. Cycles 2+ repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Trabectedin; Drug: Venetoclax
- Cohort II (BTK-intolerant) (Experimental): Patients receive trabectedin IV over 3 hours on day 1 of a 3-week cycle (cycle 1), then receive venetoclax PO QD beginning on day 1 of a 5-week cycle (cycle 2). Beginning in cycle 3, patients receive trabectedin IV over 3 hours on day 1 and venetoclax PO QD every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Trabectedin; Drug: Venetoclax

INTERVENTIONS:
Drug: Trabectedin — Given IV
  Other Names: Ecteinascidin; ecteinascidin 743; ET-743; Yondelis
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta

SUMMARY:
This phase I/Ib trial studies the best dose and side effects of trabectedin and venetoclax in treating patients with chronic lymphocytic leukemia or small lymphocytic lymphoma that is resistant or intolerant to a BTK inhibitor. Drugs used in chemotherapy, such as trabectedin and venetoclax, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate safety and tolerability, and to determine dose and schedule of trabectedin in combination with venetoclax in patients with chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) resistant or intolerant to a BTK inhibitor.

SECONDARY OBJECTIVES:

I. To determine the best response achieved by patients treated with combined trabectedin and venetoclax.

II. To determine the progression-free (PFS) and overall survival (OS) of patients treated with combined trabectedin and venetoclax.

III. To investigate the effects of trabectedin on CLL cells and on the components of the CLL microenvironment.

IV. To investigate associations between baseline characteristics (including fluorescence in situ hybridization [FISH] status, IGHV mutation status and mutations responsible for resistance to BTK inhibitors) and response to the combination of trabectedin and venetoclax.

OUTLINE: This is a dose-escalation study. Patients are assigned to 1 of 2 cohorts.

COHORT I (BTK-REFRACTORY): Patients receive venetoclax orally (PO) once daily (QD) beginning on day 1 for 5 weeks (cycle 1). Beginning in cycle 2, patients receive venetoclax PO QD and trabectedin intravenously (IV) over 3 hours on day 1. Cycles 2+ repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

COHORT II (BTK-INTOLERANT): Patients receive trabectedin IV over 3 hours on day 1 of a 3-week cycle (cycle 1), then receive venetoclax PO QD beginning on day 1 of a 5-week cycle (cycle 2). Beginning in cycle 3, patients receive trabectedin IV over 3 hours on day 1 and venetoclax PO QD every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of CLL/SLL who are progressing (based on 2018 International Workshop on Chronic Lymphocytic Leukemia [iwCLL] criteria) on or intolerant to a BTK inhibitor (BTK-inhibitor-intolerant is defined as unable to maintain on a stable and continuous dose of at least ibrutinib 140 mg/day [or acalabrutinib 100 mg/day] for at least 2 weeks due to recurrent treatment-related grade 2 or higher non-hematologic toxicity by Common Terminology Criteria for Adverse Events [CTCAE] grading)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin =< 1.0 x upper limit of normal (ULN) or =< 3 x ULN for patients with Gilbert's disease
* Creatinine clearance > 50 mL/min (calculated according to institutional standards or using Cockcroft-Gault formula)
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST) =< 2.5 x ULN
* Alkaline phosphatase (ALP) =< 2.5 x ULN
* Platelet (PLT) count >= 50,000/l, with no platelet transfusion in 2 weeks prior to registration, unless cytopenia is due to bone marrow involvement with CLL, in which case PLT count > 30,000/l, with no PLT transfusion in 2 weeks prior to registration
* Absolute neutrophil count (ANC) >= 1000/l, unless cytopenia is due to bone marrow involvement with CLL, in which case ANC > 500/l
* Creatine phosphokinase (CPK) < 2.5 x ULN
* Left ventricular ejection fraction (LVEF) assessed by multi-gated acquisition scan (MUGA) or echocardiogram within limits of normal range
* Women of childbearing potential must agree to use an effective contraception method during the study and for 60 days following the last dose of study drug. Women of non- childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy. Men who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 60 days following the last dose of study drug
* Free of prior malignancies for 2 years with exception of patients diagnosed with basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast, who are eligible even if they are currently treated or have been treated and/or diagnosed in the past 2 years prior to study enrollment. If patients have another malignancy that was treated within the last 2 years, such patients may be enrolled, if the likelihood of requiring systemic therapy for this other malignancy within 2 years is less than 20%
* Patients or their legally authorized representative must provide written informed consent

Exclusion Criteria:

* Radiotherapy or chemotherapy within 2 weeks prior to the first dose of the study drugs. Given the quick progression associated with resistance to BTK inhibitors, no limits will be placed to the use of BTK inhibitors for enrollment or initiation of treatment on this trial
* Uncontrolled active systemic infection (viral, bacterial, and fungal)
* Active, uncontrolled autoimmune phenomenon (autoimmune hemolytic anemia or immune thrombocytopenia) requiring steroid therapy with > 20 mg daily of prednisone or equivalent
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 2 months of screening, or any class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
* Patient is pregnant or breast-feeding
* Venetoclax-refractory CLL or prior treatment with trabectedin
* Malabsorption syndrome or other condition that precludes oral/enteral route of administration
* Patients who received the following within 7 days prior to first dose of venetoclax: moderate and strong CYP3A inhibitors and inducers, P-glycoprotein inhibitors, or narrow therapeutic index P-glycoprotein substrates AND patients who received the following within 3 days prior to first dose of venetoclax: grapefruit or grapefruit products, Seville oranges and star fruit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Estimated)

PRIMARY OUTCOMES:
Dose and schedule of trabectedin in combination with venetoclax | Up to 6 months post-treatment

SECONDARY OUTCOMES:
Best response | Up to 6 months post-treatment
  Will be assessed using the 2018 International Workshop on Chronic Lymphocytic Leukemia response criteria. Minimal residual disease will be evaluated by 4-color flow cytometry.
Progression free survival | From treatment initiation to disease progression or death, assessed up to 6 months post-treatment
Overall survival | From treatment initiation to death due to any cause, assessed up to 6 months post-treatment
Frequency of myeloid cells and of other immune cells | Baseline up to 6 months post-treatment
  Will be analyzed in the peripheral blood and bone marrow (if available).

CONTACTS AND LOCATIONS:
Overall Officials: William G Wierda, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org